CLINICAL TRIAL: NCT05047302
Title: Investigation of Femoropopliteal In Situ Valve Formation With the InterVene System (INFINITE-Canada)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project suspended by sponsor
Sponsor: Intervene, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN009
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Chronic Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): The goal of the BlueLeaf System is to percutaneously form one or more functional, autogenous deep venous valves and restore venous competence.
  Interventions: Device: BlueLeaf Procedure

INTERVENTIONS:
Device: BlueLeaf Procedure — The device is intended to form autogenous tissue leaflets from vein walls without the use of a permanent vascular implant.

SUMMARY:
Prospective, non-randomized, multicenter pre-market feasibility study to evaluate subjects treated with the BlueLeaf System for the treatment of symptomatic CVI of the lower extremity.

DETAILED DESCRIPTION:
STUDY DESIGN: The Study is a prospective, non-randomized study to evaluate participants treated with the BlueLeaf System for the restoration of deep venous competence for the treatment of symptomatic chronic venous insufficiency (CVI).

STUDY OVERVIEW: Potential participants who pass pre-screening and are willing to participate in the study will be asked to sign the study Informed Consent Form before any study-specific tests or procedures are performed or for any study specific evaluations not considered standard of care that need to be performed to assess eligibility.

Eligible participants may undergo the index procedure. Adverse events are assessed. All participants enrolled in the study are evaluated at pre-specified timepoints.

STUDY POPULATION: Patients with CVI and a Clinical Etiological Anatomical Pathophysiological (CEAP) classification of 4, 5, or 6.

STUDY ENROLLMENT: Up to 50 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 years of age or older;
* 2. Symptomatic CVI subjects, Clinical Etiological Anatomical Pathophysiological (CEAP) classification 4 to 6;
* 3. Failed at least 6 months of conservative therapy at some point during the course of their CVI management (symptoms not adequately resolved or patient non-compliant/unable to tolerate);
* 4. Willing and able to sign the approved informed consent form (ICF);
* 5. Willing to comply with follow-up evaluations and protocols;
* 6. Deep system venous reflux characterized by >1 second reflux time in two contiguous vein segments (vein segments defined as: proximal femoral, distal femoral, and popliteal), as assessed by DUS with patient in the standing position;
* 7. Presence of at least two potential target sites within the target vessel, which is defined as a segment within the femoral or popliteal vein that is:

  * not less than 7mm in luminal diameter, and
  * not more than 11mm in luminal diameter, and
  * at least 3cm long (two target sites in a row must be spaced at least 1cm apart), and
  * absent severe obstructive features such as thrombus, synechiae, natural valves, major tributaries (valves can be formed opposite tributaries) or severe heterogeneous fibrotic changes of the vessel wall which, in the Investigator's opinion, would preclude formation of a valve, as preliminary assessed by DUS, and then by IVUS, while the vein is under physiologically appropriate hemodynamic pressure, with IVUS being the definitive modality.
* 8. In the Investigator's opinion, the subject is a good candidate for treatment with the BlueLeaf System based on their symptoms, quality of life, anatomy, and the likelihood of benefit from continued conservative therapy.

Exclusion Criteria:

* 1. Untreated significant superficial venous incompetence within 30 days of screening which, in the opinion of the Investigator, may be the primary source of existing symptoms;
* 2. A competent vein valve in any vein segment through which the device is likely to be inserted, as assessed by DUS (<1 second reflux time) or with contrast venography (Investigator's opinion);Deep venous intervention (includes stenting) in the target limb or outflow vessels within 90 days of consent;
* 3. Deep venous intervention (includes stenting) in the target limb or outflow vessels within 90 days of consent
* 4. Significant peripheral arterial disease with an ankle-brachial index of <0.70 or with incompressible vessels;
* 5. Contraindications to all protocol specified anticoagulation options;
* 6. Known and uncontrolled hypercoagulopathy (i.e. hypercoagulopathy that cannot be adequately managed/controlled with medication);
* 7. Acute deep venous thrombosis (DVT) within 6 months of consent;
* 8. Comorbidity risks or other concerns (e.g. recent cancer) which, in the opinion of the Investigator, limit longevity or likelihood of complying with the protocol and its prescribed follow up or would preclude the patient from open surgery in the event of a complication requiring surgical intervention (e.g. severe vein laceration);
* 9. General contraindications to local, regional or general anesthesia required for the index procedure;
* 10. NYHA Class III or IV heart failure;
* 11. Active systemic infection;
* 12. Women on long-term oral contraceptives;
* 13. Subject is enrolled in another clinical study that, in the opinion of the Investigator, may conflict with this study or compromise study results;
* 14. Invasive surgical procedure within the last 90 days that in the Investigator's opinion would interfere with the study procedure or results;
* 15. History of stroke within the last 6 months;
* 16. Flow-limiting venous outflow obstruction central to the intended target sites, defined by a common femoral vein duplex exam found to have a continuous waveform without respiratory variation or a 50% or greater reduction in luminal cross-sectional area on IVUS;
* 17. Inadequate flow into or through the target vessel (Investigator's opinion);
* 18. Anatomy that does not support proper device access of the treatment vein through the ipsilateral common femoral or femoral vein;
* 19. Luminal diameter <7 mm between the vein access site and the intended treatment site, as assessed by IVUS, while the vein is under physiologically appropriate hemodynamic pressure;
* 20. A competent vein valve in any vein segment through which the device is likely to be inserted (common femoral or femoral vein)
* 21. Chronic renal insufficiency with creatinine level of ≥2mg/dL;
* 22. Hemoglobin level <9.0 mg/dL;
* 23. Platelet count <50,000 or >1,000,000 per mm3;
* 24. Total white blood cell count <3,000/mm3;
* 25. Pregnant or lactating female; positive pregnancy test, women of childbearing potential must be tested;
* 26. Non-ambulatory patients;
* 27. Patients with a history of right heart failure occurring as a consequence of, for example, biventricular failure, intrinsic pulmonary disease, chronic thromboembolic pulmonary hypertension, and other etiologies that result in elevated right-sided pressures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Venous Clinical Severity Score (VCSS) | 1 year
  A decrease in score from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Elkins, Study Director — Intervene, Inc.

IPD SHARING:
Plan to Share IPD: No